CLINICAL TRIAL: NCT05498844
Title: Adherence to Nutritional Treatment and Its Effectiveness After Myocardial Infarction Using Telemedicine Versus In-person Treatment (ADNUT)
Brief Title: Adherence to Nutritional Treatment Following MI Using Telemedicine Treatment (ADNUT)
Acronym: ADNUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ariel University (Other)
Collaborators: Sheba Medical Center (Other Government); Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Vered Kaufman Shriqui, Assistant Professor, Department of Nutrition Sciences, Ariel University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC-8448-21
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases; Acute MI
Keywords: Cardiovascular disease prevention; Digital cardiac rehabilitation; Medical Nutrition Therapy; Mediterranean diet score
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Nutrition Therapy; Counseling

STUDY DESIGN:
Intervention Model Description: In a single-blind, randomized controlled, single-center study, Individuals will be randomized to intervention or control groups by stratified randomization where the stratification will be by cardiac risk level and sex. All eligible patients fulfilling the eligibility criteria will be randomly sampled from the clinic lists. These patients will be contacted by study personnel after approval from the treating physician and asked to come for a baseline meeting and explanation of study procedures. Those meeting all inclusion criteria and willing to provide informed consent will be enrolled. A log will be kept of refusals and reasons for refusal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (Active Comparator): Control group participants will receive usual medical, physical activity, and standard in-person nutrition counseling (IPNC) on site.
  Interventions: Behavioral: Medical Nutrition Therapy (counselling)
- Intervention-remote nutrition councelling (Experimental): Intervention group participants will receive remote, web-based nutrition counseling (WBNC) in addition to the standard medical counseling and on-site physical activity.
  Interventions: Behavioral: Medical Nutrition Therapy (counselling)

INTERVENTIONS:
Behavioral: Medical Nutrition Therapy (counselling) — Participants will receive nutrition counseling to enhance adherence to the principles of the Mediterranean diet and support the achievement of adequate levels of lipid control, blood pressure and weight.

SUMMARY:
Background and aim: Cardiovascular diseases (CVDs) are the leading cause of death and disability worldwide. Although cardiac rehabilitation (CR) is an effective modality that reduces the risk for death, hospital readmissions and improves the quality of life (QoL), only a third of the patients participate in CR. The association between individual nutrients and dietary patterns such as the Mediterranean diet (MedDiet) have been shown to reduce the risk of myocardial infarction (MI) and mortality. Every 1-point increase in Mediterranean diet score is associated with a 12% decrease in mortality. Although physical activity and nutrition counseling are core components of CR, less than a third of remote CR programs provide nutrition counseling. In the current study, we aim to compare the effectiveness of remote, web-based nutrition counseling (WBNC) to standard in-person nutrition counseling (IPNC).

Methods: Patients one month or less from hospital discharge for MI, who are capable of conducting a conversation using Zoom software, will be eligible to participate. In a single-blind, controlled single-center study, a 1: 1 randomization will be performed for web-based nutrition counseling (WBNC) intervention or standard in-person nutrition counseling (IPNC). Patients from both groups will receive the usual CR program (medical follow-up and on-site physical activity). Interventions will be delivered at baseline, 45 days, and 90 days post-baseline. Follow-up assessments will be performed at 6 months. Patients will complete questionnaires for socioeconomic information, physical activity level, motivation to perform lifestyle changes, food intake, adherence to MedDiet and QoL. Anthropometric measures and handgrip strength will be obtained. Medical information, lipid profile and fasting glucose level will be obtained from patient's records. Calculated sample size: 90 patients to reject the null hypothesis (no difference in between-group adherence to MedDiet) with 80% power and a confidence interval of 95%.

Expected results: The effectiveness of WBNC on adherence to MedDiet, anthropometric measures, and Qol. Our findings will enable us to identify target populations for whom nutritional treatment using telemedicine will achieve optimal results.

Importance to Medicine: Remote nutrition counseling has the potential to increase the accessibility and participation of patients, thus reducing gaps in medical service, hospitalizations, complications, and mortality. If proven beneficial, remote treatment will also allow for continuity of treatment during emergencies and closure.

DETAILED DESCRIPTION:
Background: Cardiovascular diseases (CVDs) are the leading cause of death and disability globally (1). It has been suggested that among all modifiable risk factors for CVD, an unhealthy diet has a major contributor to morbidity and mortality from CVD (2). An extensive body of evidence has led to the development of dietary guidelines for CVD prevention (3). The Mediterranean diet has been established as a major dietary pattern for the primary prevention of CVD (4). Evolving evidence support the contribution of the Mediterranean diet to secondary CVD (4, 5). Successful cardiac rehabilitation (CR) plans are comprehensive and extensive and include medical supervision, physical activity, physiotherapy, and nutrition support. Despite being an evidence-based clinical standard, and demonstrating prevention of readmission and higher health-related quality of life (QoL)(6) referral and participation in CR are low, especially among women and older adults (7). Accessibility difficulties, group setting, non-flexible hours, long commute times, and travel costs have been identified as barriers to participating in CR programs. Remote CR programs may address accessibility barriers and may represent an alternative for certain populations, and the need to develop additional effective modalities made apparent during the COVID-19 outbreak (8). Modalities for delivering remote physical activity and cardiac monitoring have shown promising results (9) and have been implemented successfully in Israel (10). However, it remains unclear whether remotely delivered nutrition therapy is effective.

In this proposal, we suggest comparing modalities of nutrition treatment for patients in a CR program in a randomized clinical trial. We will compare existing, in-person nutrition counseling (IPNC) program to a remote, web-based nutrition counseling (WBNC) program for three months post-discharge due to Myocardial infarction (MI) and examine its effectiveness for the first six months post discharge. The primary hypothesis is that there will be greater adherence to the Mediterranean diet in participants randomly assigned to WBNC than in those randomly assigned to IPNC.

B. Study Design, including:

1. Detailed Plan of the Study; the research plan should be outlined for the whole research period requested.

   A single-blind, randomized controlled, single-center study
   1. The study population will include patients within a month within one month from hospital discharge for MI, with of cardiac risk 1-2, capable of conducting a conversation using Zoom software, in either Hebrew or English. We will exclude patients with a prognosis of one year or less due to comorbidity, patients with renal failure, or patients with hemodynamic instability, those who were already participating in a remote cardiac rehabilitation program, patients with hearing or vision impairments prevented from reasonable participation in an online call (zoom) or patients, who do not have access to a computer/smartphone.
   2. Baseline data (Time 0 - T0) Socioeconomic and lifestyle information on smoking and physical activity as well as the patient's willingness to undergo a lifestyle change will be obtained during a personal interview. Food intake will be measured using 24 H food recall, adherence to MedDiet will be measured using the I-MEDAS (11), QoL will be assessed using the SF-36 (12) . Anthropometric measures: height, weight, waist circumference and Handgrip strength (HGS) (13) will be ascertained. Information recorded from the patient chart will include blood pressure, fasting blood glucose, HbA1C, cholesterol, and smoking status (current, past, never). These measures will be recorded again 3 months at completion of the intervention (T2). Blood tests will not be performed as part of the study procedures, but records will be extracted regarding blood tests performed in routine care in the patient's HMO.
   3. Length of intervention- 3 months. Follow-up will take place immediately after the intervention (T1) and at 6 months after the intervention (T2). The main outcome variable will be adherence to MedDiet at T1 as measured by I-MEDAS (validated in the Israeli population, scores range from 1-17) (11), and the change in I-MEDAS from T0 to T1, T0 to T2, T1 to T2, and T1 to T2.
   4. The interventions will take place in Cardiac Rehabilitation Unit, Sheba Medical Center, Ramat Gan. Individuals fulfilling the eligibility criteria will receive an explanation on the study procedures. After providing written informed consent, patients will be randomly assigned to either intervention or control groups. Control group participants will receive usual medical, physical activity and standard in-person nutrition counseling (IPNC) on site. Intervention group participants will receive remote, web-based nutrition counseling (WBNC) in addition to the standard medical counseling and on-site physical activity.
2. Methods (Sample size and its justification should be included & available equipment / means)

   1. Randomization: Individuals will be randomized to intervention or control groups by stratified randomization where the stratification will be by cardiac risk level and sex. All eligible patients fulfilling the eligibility criteria will be randomly sampled from the clinic lists. These patients will be contacted by study personnel after approval from the treating physician and asked to come for a baseline meeting and explanation of study procedures. Those meeting all inclusion criteria and willing to provide informed consent will be enrolled. A log will be kept of refusals and reasons for refusal. We expect a refusal rate of 20-35%.
   2. Sample size: Assuming baseline I-MEDAS score of median (IQR) of 7(2), the study would require 35 participants per group to achieve 80% power to detect a change in mead I-MEDAS score of 2 units (e.g. to 9 (3) (assuming a larger variance in T1 and T2, T3 results than at baseline) Assuming 30% lost to follow-up, each arm will be increased to 45 per group.
   3. Statistical analysis: Due to the multilevel nature of the sampling and allocation, and presumed dependence between participants in the same clinic - multilevel analytic tools will be used. Baseline parameters including age, glucose, BP, and cholesterol measures will be compared between and among groups using multi-level linear models, while distribution of smoking and other categorical variables will be assessed using multi-level models for comparing proportions. Outcome analysis will examine median I-MEDAS across the strata and among treatment arms using linear multilevel models. We will also examine within-subject differences using repeated measures and evaluating outcomes at the three time points (T0, T1, T2 & T3).

ELIGIBILITY:
Inclusion Criteria:

* Patients within one month from hospital discharge for PTCA/MI,
* Patients with cardiac risk 1-2
* Patients capable of conducting a conversation using Zoom software
* Patients speaking either Hebrew or English

Exclusion Criteria:

* Patients with a prognosis of one year or less due to comorbidity
* Patients with renal failure or patients with hemodynamic instability
* Patients who were already participating in a remote cardiac rehabilitation program
* Patients with hearing or vision impairments are prevented from reasonable participation in an online call (zoom) or patients
* Patients who do not have access to a computer/smartphone.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-08-21 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Increase in I-MEDAS score | 6 months
  change in mean I-MEDAS score of 2 units

SECONDARY OUTCOMES:
Adherance to nutrition treatment | 6 months
  Arriving to nutrition counselling during half a year following PTCA/MI

OTHER OUTCOMES:
Muscle strength | 3 MONTHS
  As measured by hand grip

CONTACTS AND LOCATIONS:
Overall Officials: Robert Klempfner, MD, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba, Tel Hashomer Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No